CLINICAL TRIAL: NCT05777941
Title: Strength Training With Eccentric Arm-cranking in Para-athletes
Acronym: KREHA-ParAth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-06
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: eccentric; strength training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eccentric Training (Experimental): This Group will train on the KREHA for 20 Trainings
  Interventions: Other: eccentric arm-cranking training

INTERVENTIONS:
Other: eccentric arm-cranking training — Over the twenty training sessions, able-bodied participants will exercise on the KREHA device. An arm-crank has to be decelerated, which will be rotated by a prematurely defined revolution rate and training duration. During this intervention a certain power has to be applied. During the whole time of training a continous progression in power and training duration is applied.

SUMMARY:
The new training device, the eccentric arm-crank, will be examined for its training effects in athletes with a spinal cord injury (SCI) by this project. That the training device can be used in patients with paraplegia in the future, the so-called "testing of the applicability of this concept" will be carried out during this study. Fourteen volunteer, healthy athletes with SCI are first tested for their upper body performance, followed by a training phase over 20 trainings and at the end the performance data is collected again. The training intensity and duration is continuously increased during the training phase.

DETAILED DESCRIPTION:
At the beginning, the study design includes a familiarisation appointment with performance tests and training on the eccentric arm-crank device (KREHA). At least one week later, the first test sequence including a maximum strength test (bench press) and a test to determine the anaerobic performance (Wingate test) is conducted. The second test sequence takes place one to three days later. This includes a handgrip strength test, an aerobic endurance test (ramp test on the arm crank ergometer with ergospirometry) and a further familiarisation training on the KREHA. The training phase starts within two weeks after the pre-tests have been completed. There are two to a maximum of three trainings per week. These take 30 to 45 minutes and take place on the KREHA device under the supervision of the study staff. The training phase lasts a maximum of twelve weeks (20 training sessions). The first test sequence is repeated five to eight days after the last workout. The second test sequence takes place at the same time interval as in the pre-tests.

ELIGIBILITY:
Inclusion Criteria:

* male or female with traumatic or disease-related SCI
* age between 18 and 50 years
* experience in strength training
* Squad status or at least 4h per week training
* Biceps/triceps function
* healthy(study physician)
* adequately informed and confirmed per signature

Exclusion Criteria:

* findings during anamnesis of study physician
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Upper body Performance | through study completion, an average of 20 weeks
  Peak Power - maximal reached power, generated during the 30sec Wingate arm-crank test

SECONDARY OUTCOMES:
Endurance Oxygen consumption | through study completion, an average of 20 weeks
  VO2peak [ml/min/kg] - Basic Endurance test (Ergospirometry, arm-crank)
Maximal Workload | through study completion, an average of 20 weeks
  Wmax [W] - Basic Endurance test (Ergospirometry, arm-crank)
Upper body Mean Power | through study completion, an average of 20 weeks
  Mean Power [W] - Wingate Test (arm-crank)
Upper body Power - Time to Peak | through study completion, an average of 20 weeks
  Time to Peak [s] - Wingate Test (arm-crank)
Upper body Fatigue Index | through study completion, an average of 20 weeks
  Fatigue Index [%]- Wingate Test (arm-crank)
Upper body Fatigue Slope | through study completion, an average of 20 weeks
  Fatigue Slope [W/s] - Wingate Test (arm-crank)
1RM bench press | through study completion, an average of 20 weeks
  One Repetition Maximum (1RM) [kg]- bench press
Grip Strength | through study completion, an average of 20 weeks
  Maximal Force that can be generated by pressing hand towards a fist [N]
Upper Arm Circumference | through study completion, an average of 20 weeks
  Circumference of the upper arm is measured with measuring tape
Lower Arm Circumference | through study completion, an average of 20 weeks
  Circumference of the lower arm is measured with measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Ammann, MSc, Principal Investigator — SPZ
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No